CLINICAL TRIAL: NCT02939664
Title: Laparoscopic Gastric Bypass Versus Laparoscopic Banded Gastric Bypass, a Randomized Prospective Clinical Trial
Brief Title: Laparoscopic Gastric Bypass Versus Laparoscopic Banded Gastric Bypass Randomized Prospective Clinical Trial
Acronym: LGB-vs-LbGB
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Miguel J. Garcia-Oria, MD, PhD, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04252016Acta07.16
Record Dates: First submitted 2016-09-28; First posted 2016-10-20 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Morbid Obesity; Weight Loss; Postoperative Complications
Keywords: banded gastric bypass; weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Postoperative Complications | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Banded Gastric Bypass (Active Comparator): The patient will have done a laparoscopic Roux-en-Y banded (with polypropylene mesh) gastric bypass at the time of the surgical procedure.
  Interventions: Device: Banded (with polypropylene mesh) gastric bypass
- Gastric Bypass. (Active Comparator): The patient will have done a Laparoscopic Roux-en-Y gastric bypass at the time of the surgical procedure
  Interventions: Procedure: Gastric bypass

INTERVENTIONS:
Device: Banded (with polypropylene mesh) gastric bypass — The patient will be submitted to a Laparoscopic Roux-en-Y banded gastric bypass at the time of the operation, with a polypropylene mesh around the gastric pouch.
  Other Names: Laparoscopic banded gastric bypass; Laparoscopic Roux-en-Y banded gastric bypass; Laparoscopic Banded Roux-en-Y gastric bypass
  Arms: Banded Gastric Bypass
Procedure: Gastric bypass — In this case a simplified conventional gastric bypass will be performed
  Other Names: Laparoscopic Gastric bypass
  Arms: Gastric Bypass.

SUMMARY:
This study try to identify differences in length of operation, weight loss and complications, between two different bariatric surgical techniques, the laparoscopic Roux-en-Y gastric bypass and the laparoscopic Roux-en-Y banded gastric bypass. The study will be conducted in a Spanish public health system hospital. The patients of the trial will have the preoperative studies, hospital treatment during the admission, postoperative treatment and follow up as any other patient included in the hospital bariatric surgery program. The study cases will have placed around the gastric pouch a band of polypropylene mesh, and will be randomly choose between the participants.

Patients will be randomized in a 5/3 (study/control) ratio.

DETAILED DESCRIPTION:
One group of patients of the study will have done the simplified laparoscopic gastric bypass, with a vertical gastric pouch of about 20 ml, a 150 cm Roux-en-Y limb constructed in an antegastric antecolic fashion, and a biliary limb of 100 cm. Anastomosis will be done with endoscopic surgical linear stapler, closing the apertures with continuous absorbable running sutures. The Petersen space and the mesenteric defect will be closed with non-absorbable sutures.

The other group of patients will have performed the laparoscopic Roux-en-Y banded gastric bypass. This technique is identical to the one performed in the other group, but differs in that a polypropylene mesh (10x65 mm) is placed 15 mm proximal to the anastomosis around the gastric pouch, and the gastric pouch is about 15 mm longer.

The investigators randomly assigned 50 patients to the study group (Laparoscopic Roux-en-Y banded gastric bypass) and 30 to the control group (Laparoscopic Roux-en-Y gastric bypass) , n=80, and were also blinded to the surgeon until surgery.

One of the methods is basically the same than the other, but for the placement of the polypropylene mesh around the gastric pouch above the anastomosis, and patient series with Laparoscopic Roux-en-Y banded gastric bypass showed long term better weight loss than other series with not banded gastric bypass, thus it is expected a difference in long term weight loss between groups.

Fisher Test will be used for the statistical analysis, assuming a risk of 0.05 and a statistical power of 90%.

Sample size is calculated considering bibliographic long term weight loss in both groups, which is 82% in the banded group versus 63% in the not banded group. Thus sample size (n): 67, and adjust by loss sample size: 79 (10% expected loss ratio), not being necessary a 1: 1 ratio between cases and controls and requiring no more than 25 controls, A sample size of 50 cases and 30 controls, total n = 80, will be used.

The method of randomization was concealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* criteria for bariatric surgery published in 1991 for the National Institutes of Health of the USA.
* Body mass index (BMI)> 40 and <55 kg/m2
* Obesity for more than 5 years of evolution
* Fail in medical supervised weight loss program
* patient knowing of the mechanism of weight loss after surgery and agreement to collaborate with medical recommendations, diet, medical treatment, as well as the visit established in the follow up program
* patient accepting that surgery objective is not to achieve the ideal weight.
* signed specific informed consent
* women will agree in avoid gestation during one year after surgery

Exclusion Criteria:

* Patients unable to sign the informed consent form because of a mental disorder.
* endocrine diseases causing obesity
* unstable mental disorder, evaluated for a psychiatry MD.
* high anesthetic risk making surgery too risky.
* Malignant neoplasm
* Inflammatory bowel disease
* Severe liver disease
* Digestive disease that makes unwise the bypass technique (mainly gastric illness that may required upper endoscopy for control)
* abdominal wall hernias
* Symptomatic biliary pathology that requires cholechistectomy at the same time of the bariatric surgery
* any known pathology that requieres or recomend simultaneous surgery at the time of the bariatric surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2034-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Change from operation date, in excess weight loss at 10 years | 10 years
  % of excess weight loss at 10 years
Postoperative complications at 10 years | 10 years
  Number of participants with adverse events (surgical complications) and/or abnormal Laboratory values that are related to treatment

SECONDARY OUTCOMES:
Excess weight loss at 5 years | 5 years
  % of excess weight loss at 5 years
Total Hospital cost at 3 months | up to 3 months
  Total hospital expenses during admission for the surgery and 3 months after the operation.
Postoperative complications 1 year | 1 year
  Number of participants with adverse events (surgical complications)
Postoperative complications 2 years | 2 years
  Number of participants with adverse events (surgical complications)
Postoperative complications 3 years | 3 years
  Number of participants with adverse events (surgical complications)
Postoperative complications 5 years | 5 years
  Number of participants with adverse events (surgical complications)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel J Garcia-Oria, MD PhD FACS, Study Chair — General Surgery Department. Hospital Universitario Puerta de Hierro; Miguel J Garcia-Oria, MD PhD, Study Director — Servicio de Cirugía General. Hospital Universitario Puerta de Hierro Majadahonda
Locations (1):
- Servicio de Cirugía General. Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
We will publish the results of the study in a surgical journal

REFERENCES:
- [Background] Arceo-Olaiz R, Espana-Gomez MN, Montalvo-Hernandez J, Velazquez-Fernandez D, Pantoja JP, Herrera MF. Maximal weight loss after banded and unbanded laparoscopic Roux-en-Y gastric bypass: a randomized controlled trial. Surg Obes Relat Dis. 2008 Jul-Aug;4(4):507-11. doi: 10.1016/j.soard.2007.11.006. Epub 2008 Jan 28. PMID 18226982
- [Background] Bessler M, Daud A, Kim T, DiGiorgi M. Prospective randomized trial of banded versus nonbanded gastric bypass for the super obese: early results. Surg Obes Relat Dis. 2007 Jul-Aug;3(4):480-4; discussion 484-5. doi: 10.1016/j.soard.2007.01.010. Epub 2007 Jun 4. PMID 17544335
- [Background] Buchwald H, Buchwald JN, McGlennon TW. Systematic review and meta-analysis of medium-term outcomes after banded Roux-en-Y gastric bypass. Obes Surg. 2014 Sep;24(9):1536-51. doi: 10.1007/s11695-014-1311-1. PMID 25001288
- [Background] Capella JF, Capella RF. An assessment of vertical banded gastroplasty-Roux-en-Y gastric bypass for the treatment of morbid obesity. Am J Surg. 2002 Feb;183(2):117-23. doi: 10.1016/s0002-9610(01)00871-6. PMID 11918873
- [Background] Capella JF, Capella RF. The weight reduction operation of choice: vertical banded gastroplasty or gastric bypass? Am J Surg. 1996 Jan;171(1):74-9. doi: 10.1016/S0002-9610(99)80077-4. PMID 8554155
- [Background] Mahawar KK, Parikh C, Carr WR, Jennings N, Balupuri S, Small PK. Primary banded Roux-en-Y gastric bypass: a systematic review. Obes Surg. 2014 Oct;24(10):1771-92. doi: 10.1007/s11695-014-1346-3. PMID 24968745
- [Background] Rasera I Jr, Coelho TH, Ravelli MN, Oliveira MR, Leite CV, Naresse LE, Henry MA. A Comparative, Prospective and Randomized Evaluation of Roux-en-Y Gastric Bypass With and Without the Silastic Ring: A 2-Year Follow Up Preliminary Report on Weight Loss and Quality of Life. Obes Surg. 2016 Apr;26(4):762-8. doi: 10.1007/s11695-015-1851-z. PMID 26314349
- [Background] Zarate X, Arceo-Olaiz R, Montalvo Hernandez J, Garcia-Garcia E, Pablo Pantoja J, Herrera MF. Long-term results of a randomized trial comparing banded versus standard laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2013 May-Jun;9(3):395-7. doi: 10.1016/j.soard.2012.09.009. Epub 2012 Oct 3. PMID 23260801